CLINICAL TRIAL: NCT01947153
Title: Two-way Crossover Study in Healthy Male and Female Subjects to Evaluate the Bioequivalence of Jentadueto® (Two Fixed Dose Combination Tablets of Linagliptin 2.5 mg and Metformin 500 mg) Compared With the Free Combination of Linagliptin 5 mg and Metformin 1000 mg Tablets Under Fasting Conditions.
Brief Title: Two-way Crossover Study in Healthy Male and Female Subjects to Evaluate the Bioequivalence of Jentadueto®.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.21
Record Dates: First submitted 2013-09-18; First posted 2013-09-20 (Estimated); Results first posted 2015-02-25 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin; Linagliptin

ARMS (2):
- Fixed dose combination (Experimental): Linagliptin/Metformin
  Interventions: Drug: Linagliptin; Drug: Metformin
- Free combination (Experimental): Linagliptin and Metformin
  Interventions: Drug: Metformin; Drug: Linagliptin

INTERVENTIONS:
Drug: Metformin — Free combination
  Arms: Free combination
Drug: Linagliptin — Fixed dose combination
  Arms: Fixed dose combination
Drug: Metformin — Combination
  Arms: Fixed dose combination
Drug: Linagliptin — Free combination
  Arms: Free combination

SUMMARY:
The objective of the current study is to demonstrate bioequivalence of two 2.5 mg linagliptin/500 mg metformin fixed dose combination tablets compared to the free combination of the linagliptin 5 mg and metformin 1000 mg in healthy male and female volunteers.

ELIGIBILITY:
Inclusion criteria:

* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation
* Healthy males and females according to the following criteria:

Based upon a complete medical history, including physical examination, vital signs (BP, PR), 12-lead ECG and clinical laboratory tests (haematology, clinical chemistry and urinalysis).

* Age 18 to 45 years (incl.)
* Body mass index by Quetelet between 18.50 to 24.99 kg/m2 (incl.)
* Female subjects of childbearing potential who agree on using double-barrier contraception during the study. If a female is postmenopausal (no menses for at least 2 years) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) she will be exempt from the requirement. In case of using oral contraceptives, these should be withdrawn at least 2 months before the first drug dosing.
* Male subjects who agree on using effective contraception during the study (barrier contraceptive methods)

Exclusion criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any laboratory value outside the reference range that is of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Positive results of blood tests for infections (HIV, syphilis, hepatitis B or C)
* A positive urine drug screening test at screening and on admission to the trial site in each treatment period.
* A positive alcohol breath test at screening and on admission to the trial site in each treatment period.
* Surgery of the gastrointestinal tract (except appendectomy)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1288.21.1 Boehringer Ingelheim Investigational Site, Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- Fixed Dose Combination First, Then Free Combination: 5 mg linagliptin / 1000mg metformin given as two 2.5mg linagliptin / 500mg metformin fixed dose combination (FDC) tablets first; then free combination: one 5mg linagliptin tablet and one 1000mg metformin tablet
- Free Combination First, Then Fixed Dose Combination: Free combination: one 5mg linagliptin tablet and one 1000mg metformin tablet first; then 5 mg linagliptin / 1000mg metformin given as two 2.5mg linagliptin / 500mg metformin fixed dose combination (FDC) tablets
Period: Test Period 1
Arm/Group | Fixed Dose Combination First, Then Free Combination | Free Combination First, Then Fixed Dose Combination
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Test Period 2
Arm/Group | Fixed Dose Combination First, Then Free Combination | Free Combination First, Then Fixed Dose Combination
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): includes all subjects who had been dispensed study medication and were documented to have taken at least 1 dose of study medication.
Groups:
- All Subjects: All subjects treated with 5 mg linagliptin / 1000 mg metformin as fixed dose combination or as free dose combination.
Arm/Group | All Subjects
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Linagliptin: AUC 0-72 (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to 72 Hours)
Description: Linagliptin:
  AUC 0-72 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 hours)
Time Frame: 2 hours (h) before drug administration and 20 minutes (min), 40min, 1h, 1h 30min, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h and 72h after drug administration
Population: subject set for the evaluation of pharmacokinetic endpoints of linagliptin (PKS-L): includes all subjects of the TS who provided at least 1 observation for at least 1 primary endpoint for linagliptin and had no important protocol violations with respect to the statistical evaluation of pharmacokinetic endpoints of linagliptin
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Fixed Dose Combination: Linagliptin/Metformin
  Linagliptin: Fixed dose combination: 2x 2.5mg Metformin: Combination: 500mg
- Free Combination: Linagliptin and Metformin
  Metformin: Free combination 5mg Linagliptin: Free combination 1000mg
Arm/Group | Fixed Dose Combination | Free Combination
Number analyzed (Participants) | 36 | 34
nmol*h/L | 293 (23.4) | 288 (22.9)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Free Combination; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p < 0.0001, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 102.92, 90% CI 2-sided [98.370 to 107.688], Standard Error of Mean 1.027 — The geometric mean ratio is calculated as the geometric mean of 'Fixed dose combination' divided by the geometric mean of 'Free combination '

2. Primary Outcome: Metformin: AUC0-tz (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point)
Description: Metformin:
  AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point)
Time Frame: as for outcome 1
Population: The subject set for the evaluation of pharmacokinetic endpoints of metformin (PKS-M): includes all subjects of the TS who provided at least 1 observation for at least 1 primary endpoint for metformin and had no important protocol violations with respect to the statistical evaluation of pharmacokinetic endpoints of metformin
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Fixed Dose Combination | Free Combination
Number analyzed (Participants) | 36 | 34
ng*h/mL | 13000 (27.3) | 12100 (24.2)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Free Combination; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p < 0.0001, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 105.14, 90% CI 2-sided [99.645 to 110.941], Standard Error of Mean 1.032 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Linagliptin: Cmax (Maximum Measured Concentration of the Analyte in Plasma)
Description: Linagliptin:
  Cmax (maximum measured concentration of the analyte in plasma)
Time Frame: as for outcome 1
Population: PKS-L: includes all subjects of the TS who provided at least 1 observation for at least 1 primary endpoint for linagliptin and had no important protocol violations with respect to the statistical evaluation of pharmacokinetic endpoints of linagliptin
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Fixed Dose Combination | Free Combination
Number analyzed (Participants) | 36 | 34
nmol/L | 10.3 (36.4) | 9.57 (36.2)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Free Combination; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p = 0.0014, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 109.05, 90% CI 2-sided [98.299 to 120.968], Standard Error of Mean 1.063 — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Metformin: Cmax (Maximum Measured Concentration of the Analyte in Plasma)
Description: Metformin:
  Cmax (maximum measured concentration of the analyte in plasma)
Time Frame: as for outcome 1
Population: PKS-M: includes all subjects of the TS who provided at least 1 observation for at least 1 primary endpoint for metformin and had no important protocol violations with respect to the statistical evaluation of pharmacokinetic endpoints of metformin
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Fixed Dose Combination | Free Combination
Number analyzed (Participants) | 36 | 34
ng/mL | 1840 (28.2) | 1700 (27.0)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Free Combination; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p < 0.0001, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 105.81, 90% CI 2-sided [98.471 to 113.692], Standard Error of Mean 1.043 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Linagliptin: AUC 0-inf (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: Linagliptin:
  AUC 0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Fixed Dose Combination | Free Combination
Number analyzed (Participants) | 36 | 34
nmol*h/L | 467 (25.8) | 479 (29.5)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Free Combination; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p < 0.0001, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 98.48, 90% CI 2-sided [92.177 to 105.208], Standard Error of Mean 1.040 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Metformin: AUC 0-inf (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity)
Description: Metformin:
  AUC 0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Fixed Dose Combination | Free Combination
Number analyzed (Participants) | 36 | 34
ng*h/mL | 13400 (26.8) | 12500 (24.1)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Free Combination; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p < 0.0001, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 104.62, 90% CI 2-sided [99.274 to 110.254], Standard Error of Mean 1.031 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Linagliptin: AUC 0-tz (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point)
Description: Linagliptin:
  AUC 0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point)
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Fixed Dose Combination | Free Combination
Number analyzed (Participants) | 36 | 34
nmol*h/L | 293 (23.4) | 288 (22.9)
Statistical Analysis 1: Comparison: Fixed Dose Combination vs Free Combination; Test type: Non-Inferiority or Equivalence — Bioequivalence test; p < 0.0001, ANOVA — The p-value relates to the null hypothesis of non-equivalence; Geometric mean ratio = 102.92, 90% CI 2-sided [98.370 to 107.688], Standard Error of Mean 1.027 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first study drug administration until 30±2 days after the last study drug administration
Arm/Group | Fixed Dose Combination | Free Combination
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/36 | 4/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Dose Combination (N=36) | Free Combination (N=36)
Headache (Nervous system disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.